CLINICAL TRIAL: NCT03772886
Title: Reducing Cesarean Delivery Rate in Obese Patients Using the Peanut Ball: A Randomized Control Trial
Brief Title: Reducing Cesarean Delivery Rate in Obese Patients Using the Peanut Ball
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to complete enrollment
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Awathif Dhanya Mackeen, Division of Maternal-Fetal Medicine, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0613
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Obesity; Cesarean Section
Keywords: Peanut Ball
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peanut Ball Arm (Experimental): Study participants randomized to the Peanut Ball Arm will have the peanut ball placed during labor. Study participants will be required to use the peanut ball for a minimum of 30 minutes of each hour until they reach complete dilation. Peanut ball use time will be noted in the patient's chart.
  Interventions: Device: Peanut Ball
- Control Arm (No Intervention): Study participants randomized to the Control Arm will labor without the peanut ball.

INTERVENTIONS:
Device: Peanut Ball — A peanut shaped exercise ball.
  Arms: Peanut Ball Arm

SUMMARY:
This study aims to determine if using the peanut ball during labor reduces the cesarean delivery rate when compared to normal intrapartum management (no peanut ball) in the obese patient population.

DETAILED DESCRIPTION:
Currently at Geisinger Medical Center Danville, use of the peanut ball is at the discretion of attending or resident physicians, or obstetric nurses on the Labor and delivery team for the day. Despite the common use of this labor adjuvant tool, a well-designed prospective study is necessary to investigate if the peanut ball provides any benefit during the labor process for the obese gravida. If this simple tool is shown to reduce the rate of cesarean delivery, then hospital protocols could be changed to ensure its use during labor. This has the potential to decrease the rate of cesarean delivery in the most vulnerable patient population. The investigators propose a randomized controlled trial (RCT) to determine if using the peanut ball during labor provides a reduction in the cesarean delivery rate in the obese patient population. The investigators will compare cesarean delivery rates in patients using the peanut ball to patients receiving routine intrapartum management without the use of the peanut ball. Singleton pregnancies complicated by obesity, defined by pre-pregnancy BMI > 30kg/m2, will be included.

Study participants will be randomized to one of the two study arms. The peanut ball arm (also referred to as study arm 1) will be managed according to the parameters specified for use of the peanut ball. The participants in the Control arm (also referred to as study arm 2) will be managed according to the standard intrapartum management as defined by Geisinger's Labor & Delivery protocol and per the OB providers. The objective of the study is to determine if use of the peanut ball during labor reduces the cesarean delivery rate in the obese patient population. Secondary outcomes of interest include rate of cervical dilation, rate of operative deliveries, fetal position (occiput anterior vs. occiput posterior) at complete dilation (10 cm), and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Admitted for delivery
* Pre-pregnancy BMI > 30kg/m2
* Planned vaginal delivery at Geisinger Medical Center (GMC)
* Gestational age > 37 weeks 0 days
* Singleton pregnancy
* Cephalic presentation
* English speaking

Exclusion Criteria:

* Pre-pregnancy BMI < 30kg/m2
* Contraindication to vaginal delivery
* Planned cesarean delivery (i.e., an elective primary or repeat cesarean delivery)
* Gestational age < 37 weeks 0 days
* Multifetal gestation
* Intrauterine fetal demise
* Non-English speaking
* Greater than 9cm at the time of randomization

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Cesarean Delivery Rate | Delivery
  Number of vaginal deliveries vs. Number of cesarean deliveries

SECONDARY OUTCOMES:
Rate of Cervical Dilation | Randomization until complete dilation (10cm)
  The average amount of cervical dilation (cm) per hour compared between the two groups (peanut ball vs. no peanut ball).
Type of Vaginal Delivery | Delivery
  Number of spontaneous vaginal deliveries vs Number of forceps assisted vaginal deliveries vs Number of vacuum assisted vaginal deliveries.
Fetal Position | Complete Dilation (10cm)
  Occiput anterior versus occiput posterior versus occiput transverse

OTHER OUTCOMES:
Patient Satisfaction Survey | Postpartum Day One
  Evaluating overall patient satisfaction during labor course

CONTACTS AND LOCATIONS:
Overall Officials: Awathif D Mackeen, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Medical Center, Danville, Pennsylvania, United States